CLINICAL TRIAL: NCT00346255
Title: A Phase I Study to Assess The Safety and Pharmacokinetics of BB-10901 (huN901-DM1) Given as an Intravenous Infusion Weekly for Two Consecutive Weeks Every Three Weeks to Subjects With Relapsed and Relapsed Refractory CD56-Positive Multiple Myeloma
Brief Title: BB-10901 in Treating Patients With Relapsed and/or Refractory Multiple Myeloma
Acronym: IMGN901
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoGen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000491241; IMMUNO-003; DFCI-05031; NCT00625508 (obsolete NCT alias)
Record Dates: First submitted 2006-06-28; First posted 2006-06-29 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Myeloma
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — lorvotuzumab mertansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: BB-10901 — dose escalation study, doses will vary per cohort. patients will receive an IV infusion weekly for two weeks every three weeks.
  Other Names: IMGN901

SUMMARY:
RATIONALE: Monoclonal antibodies, such as BB-10901, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them.

PURPOSE: This phase I trial is studying the side effects and best dose of BB-10901 in treating patients with relapsed and/or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity and the maximum tolerated dose of BB-10901 in patients with relapsed and/or refractory CD56-positive multiple myeloma.

Secondary

* To determine the qualitative and quantitative toxicities of BB-10901 administered on this schedule.
* To evaluate the pharmacokinetics of BB-10901.
* To recommend a dose for Phase II clinical studies with BB-10901 given on this specific regimen.
* To observe any evidence of anti-tumor activity with BB-10901.

Objectives of MTD Expansion Cohort

* To evaluate response rate including overall response rate (ORR) and complete response rate (CRR), and duration of response (DOR).
* To further assess time to progression (TTP), progression free survival (PFS), and overall survival (OS).

OUTLINE: This is an open-label, non-randomized, dose-escalation, multicenter study.

Patients receive BB-10901 IV over 1-2 hours on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of BB-10901 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Up to 40 patients are treated at the MTD.

After completion of study treatment, patients are followed for short term follow-up and long term (up to 3 years) survival status.

PROJECTED ACCRUAL: A total of 80 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed multiple myeloma
* Relapsed or relapsed/refractory disease

  * Failed ≥ 1 prior therapy for multiple myeloma
  * Once the MTD is defined, only patients who have received at least 1 but equal or less than 6 prior chemotherapy regimens will be enrolled at this dose level
* CD56-positive disease confirmed by immunohistochemistry or flow cytometry

PATIENT CHARACTERISTICS:

* ECOG (Zubrod) performance status 0-2
* Life expectancy ≥ 12 weeks
* Platelet count ≥ 75,000/mm^3
* Absolute neutrophil count > 1,000/mm^3
* Hemoglobin ≥ 8.5 g/dL
* AST and ALT ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Amylase and lipase within normal limits
* Creatinine ≤ 2 mg/dL
* Left ventricular ejection fraction ≥ lower limit of normal on MUGA or ECHO
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy ≥ grade 3 or painful grade 2 neuropathy
* No significant cardiac disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * Unstable angina
  * Uncontrolled congestive heart failure
  * Uncontrolled hypertension (i.e., recurrent or persistent increases in systolic blood pressure ≥ 180 mm Hg or diastolic blood pressure ≥ 110 mm Hg)
  * Uncontrolled cardiac arrhythmias
  * Cardiac toxicity ≥ grade 3 after prior chemotherapy
* No history of multiple sclerosis or other demyelinating disease
* No hemorrhagic or ischemic stroke within the past 6 months
* No Eaton-Lambert syndrome (para-neoplastic syndrome)
* No CNS injury with residual neurological deficit (other than peripheral neuropathy ≤ grade 2)
* No other malignancy within the past 3 years except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, in situ breast cancer, or in situ prostate cancer
* No clinically relevant active infection, including active hepatitis B or C infection or HIV infection
* No other condition or disease, including laboratory abnormalities, that, in the opinion of the investigator, may preclude study treatment
* No known recent biochemical or clinical evidence of pancreatitis or extensive metastatic disease involving the pancreas

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* At least 4 weeks since prior radiotherapy
* At least 4 weeks since prior major surgery (except placement of a vascular access device or tumor biopsies)
* More than 4 weeks since prior investigational agents
* At least 2 weeks since prior antineoplastic therapy with biological agents
* No prior hypersensitivity to monoclonal antibody therapy
* No other concurrent investigational agents
* No concurrent corticosteroids (except as indicated for other medical conditions [< 10 mg prednisone or equivalent]; as pre-medication for administration of certain medications or blood products [≤ 100 mg hydrocortisone]; or for treatment of infusion reactions)

  * Concurrent topical steroids allowed
* No other concurrent antineoplastic treatment (e.g., chemotherapy, radiotherapy, or biological agents)
* Concurrent bisphosphonates allowed provided patient began bisphosphonates before study entry and is maintained on a stable dose during study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2005-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity | through cycle 1
Maximum tolerated dose | for the duration of the study

SECONDARY OUTCOMES:
Qualitative and quantitative toxicities | for the duration of the study
Pharmacokinetics | for the duration of the study
Anti-tumor activity including overall response rate, time to progression and survival | for the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Asher Alban Akmal Chanan-Khan,, M.D., Principal Investigator — Roswell Park Cancer Institute
Locations (8):
- United States (5):
  - Cedars-Sinai Outpatient Cancer Center, Los Angeles, California
  - UCSF, San Francisco, California
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - St. Vincent's Comprehensive Cancer Center - Manhattan, New York, New York
- Argentina (3):
  - Juan Domingo Peron 1500 - (B1629AHJ) Pilar, Buenos Aires, Buenos Aires
  - Gascon 450 - (C1181ACH), Buenos Aires, Buenos Aires F.D.
  - Av. Naciones Unidas 346. (X5016KEH)-Barrio Parque Velez Sarfield, Córdoba, Córdoba Province